CLINICAL TRIAL: NCT04356222
Title: Efficacy and Safety of Durvalumab Combined With Intrathecal Chemotherapy in Non-Small Cell Lung Cancer With Leptomeningeal Metastasis
Brief Title: Efficacy and Safety of Durvalumab in Non-Small Cell Lung Cancer With Leptomeningeal Metastasis
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Hui Bu (Other)
Responsible Party: Sponsor-Investigator, Hui Bu, Study Principal Investigator, Hebei Medical University
Organization: Hebei Medical University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BH 004
Record Dates: First submitted 2020-04-18; First posted 2020-04-22 (Actual); Last update posted 2020-05-27 (Actual); Status verified 2020-05

CONDITIONS: Leptomeningeal Metastasis; Durvalumab
Keywords: Leptomeningeal Metastasis; Durvalumab; Intrathecal chemotherapy
MeSH Terms: conditions — Meningeal Carcinomatosis | interventions — durvalumab; Methotrexate

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Leptomeningeal Metastasis (Experimental): Durvalumab + Intrathecal chemotherapy
  Interventions: Drug: Durvalumab; Drug: methotrexate

INTERVENTIONS:
Drug: Durvalumab — Intravenous infusion once every two weeks ,once 10mg/kg.
Drug: methotrexate — Intrathecal chemotherapy specified dose on specified days

SUMMARY:
The purpose of this study is to observe the clinical efficacy and safety of Durvalumab combined with intrathecal chemotherapy in non-small cell lung cancer with leptomeningeal metastasis

ELIGIBILITY:
Inclusion Criteria:

1. Male and Female age 18 or more
2. Pathologically proven non-small cell lung cancer
3. MRI(Magnetic Resonance Imaging,MRI) imaging findings or the detection of malignant cells in cerebrospinal fluid
4. Patients have the ability to understand and the willingness to sign a written informed consent document.

Exclusion Criteria:

1. KPS score <60
2. History of autoimmune diseases
3. With severe hepatic and renal dysfunction
4. Has a history of (non-infectious) pneumonitis that required steroids

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2020-06 (Estimated); Primary Completion 2023-06 (Estimated); Study Completion 2023-06 (Estimated)

PRIMARY OUTCOMES:
overall survival (OS) | 36 months
  OS was defined as the time between the start of treatment to the date of death or date participant was last known to be alive
Neurological Progression Free Survival(NPFS) | 36 months
  NPFS was defined as the time between the start of treatment until central nervous system metastase progression or death due to any cause
The incidence of adverse reactions | 36 months
  In accordance with the standard of CTCAE, an assessment will be assessed every 4 weeks

SECONDARY OUTCOMES:
Progression Free Survival(PFS) | 36 months
  NPFS was defined as the time between the start of treatment to the date of the first documented tumor progression as determined by investigators per RECIST 1.1,or death due to any cause
Objective response rate (ORR) | 36 months
  Investigator assessed ORR was defined as the number of subjects whose best objective response (OOR) was a confirmed complete response (CR) or confirmed partial response (PR)
Neurological assessment | 36 months
  In accordance with the standard of Response Assessment in Neuro-Oncology(RANO) Neurological Assessment group.The maximum value is 29 and the minimum value is 0.The higher scores mean a worse outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Hui Bu, Principal Investigator — The Second Hospital of Hebei Medical University